CLINICAL TRIAL: NCT01018667
Title: The ADOPT Trial (Assessment of Efficacies of Cardiac Resynchronization Therapies (CRT-P/D) for Heart Failure Patients in China): Rationale, Design and End-points
Brief Title: Assessment of Efficacies of Cardiac Resynchronization Therapies (CRT-P/D) for Heart Failure Patients in China
Acronym: ADOPT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Dr. Wang HC/Department of Cardiology, xijing hospital, Department of Cardiology, xijing hospital
Other Study IDs: Xijing-1
Record Dates: First submitted 2009-11-22; First posted 2009-11-25 (Estimated); Last update posted 2010-07-23 (Estimated); Status verified 2010-06

CONDITIONS: Heart Failure
Keywords: Heart Failure; clinical trial; biventricular pacing; cardiac device
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- CRT group
- OPT group

SUMMARY:
The ADOPT study is a prospective, nested case-controlled and open label clinical trial. About 40 centers across China participate in this study with a planned 800 Chinese cases enrollment. All patients will receive optimal medical treatment. Patients who have successful CRT-P/D implant will be assigned to CRT group. According to the baseline evaluation, matched cases will be selected from the enrolled OPT(optimal medical treatment) alone group (Group for Selection). After successful match, the cases in Group for Selection enters into follow-up and become control group. The unmatched cases in the Group for Selection will be removed. If patients agree, after re-evaluation of the baseline situation, she or he may enter into Group for Selection again. Since patients know she/he already have a device implant and the examiners are aware of the grouping of the patients after seeing the incision scar and post-implant electrocardiogram, this study is open-label designed, however the executive committee will be kept blind when making event-adjudication. Prospectively defined primary end points for the study include combined all-cause mortality and hospitalizations. A variety of secondary end points will further define the efficacy and mechanism(s) of action of cardiac resynchronization in heart failure. The last date of the study shall be the day after 24 months of follow-up of the last enrolled patient. All cases collection complete in 2010 and study result will be reported in 2012.

ELIGIBILITY:
Inclusion Criteria:

Heart failure patients who must meet all criteria:1.ischemic or nonischemic cardiomyopathy;2.NYHA classes III-IV despite OPT;3.normal sinus rhythm;4.LVEF≤35%;5.LV end-diastolic diameter≥55mm;and 6.Wide QRS complex≥120ms.

Exclusion Criteria:

1.Potentially reversible forms of cardiomyopathy;2.Cardiac surgery, percutaneous coronary intervention, cardiomyoplasty, myocardial infarction, unstable or severe angina or stroke within 6 weeks before randomization;3.In-patients requiring continuous intravenous therapy for heart failure;4.Life expectancy<1 year for disease unrelated to heart failure;5.Mechanical tricuspid valve;6.Anticipated problem with compliance;7.Participation in another trial;8.Age<18 years old;9.Women who are pregnant or not using medically acceptable birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: About eight hundred patients will be enrolled in this study at more than 40 centers in the China. To participate in the study, patients must meet the Guideline for cardiac resynchronization therapy in patients with chronic heart failure in China.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2008-10; Primary Completion 2011-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology,xijing hospital, Xi'an, Shaanxi, China